CLINICAL TRIAL: NCT07272278
Title: Prospective Clinical Study on the Clinical Efficacy and Prognostic Outcome of ICS/LABA Combined With Liqin Zhike Formula in the Treatment of Cough Variant Asthma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-1288
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Asthma
Keywords: symptom recurrence rate; cough; ICS/LABA; Traditional Chinese Medicine (TCM) treatment; Liqin Zhike Formula
MeSH Terms: conditions — Asthma; Cough

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Western Medicine Therapy Group (Active Comparator): CVA patients receive ICS/LABA treatment
  Interventions: Drug: ICS+LABA
- Integrated Chinese and Western Medicine Therapy Group (Experimental): CVA patients receive ICS/LABA treatment and Chinese medicine treatment (Liqin Zhike Formula)
  Interventions: Drug: ICS+LABA; Drug: Chinese Medicine Formula

INTERVENTIONS:
Drug: ICS+LABA — CVA patients receive ICS/LABA treatment
Drug: Chinese Medicine Formula — CVA patients receive ICS/LABA + Liqin Zhike Formula treatment
  Arms: Integrated Chinese and Western Medicine Therapy Group

SUMMARY:
To investigate the impact of the combination of ICS/LABA and Liqin Zhike Formula on the clinical efficacy and prognostic outcomes of cough variant asthma.

DETAILED DESCRIPTION:
A total of 236 patients with cough variant asthma were enrolled and randomly assigned in a 1:1 ratio. Among them, 118 patients were allocated to the Western medicine treatment group and received ICS/LABA + conventional therapy, while the other 118 patients were assigned to the integrated Chinese and Western medicine treatment group and received ICS/LABA + Liqin Zhike Formula. The treatment intervention period for both groups was 2 months, followed by a 12-month drug-discontinuation follow-up. During the 12-month follow-up period, symptom recurrence rate, asthma symptom remission rate, and adverse reactions were observed. The primary study endpoint was the symptom recurrence rate in patients with cough variant asthma during the 12-month follow-up. The secondary study endpoints were the asthma symptom remission rate and adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

- The subject voluntarily participates in this study, complies with the study regulations, understands, agrees to, and cooperates with the required examinations, adheres to the follow-up plan, and voluntarily signs the written informed consent form.

Outpatients, with age between 18 and 70 years old (inclusive).

Newly diagnosed with Cough Variant Asthma (CVA) based on clinical symptoms and pulmonary function results, according to the Chinese Bronchial Asthma Prevention and Treatment Guidelines (2024 Edition) and the Guidelines for the Diagnosis and Treatment of Cough (2021 Edition). This involves chronic cough (lasting over 8 weeks) without accompanying wheezing symptoms or signs, often occurring at night and/or early morning and worsening after exercise. All patients must meet at least one of the following pulmonary function criteria, indicating variable airflow limitation, as objective evidence for asthma diagnosis:

Objective Tests for Variable Airflow Limitation:

1. Positive bronchodilator test: An increase in Forced Expiratory Volume in one second (FEV1) of ≥12% and an absolute increase in FEV1 of ≥200 ml after inhalation of a bronchodilator; OR an increase in FEV1 of ≥12% compared to baseline and an absolute increase of ≥200 ml after 4 weeks of anti-inflammatory treatment containing Inhaled Corticosteroids (ICS) (excluding respiratory infections).
2. Positive bronchial provocation test: Commonly used inhaled agents are methacholine or histamine. A positive result is typically defined as a ≥20% decrease in FEV1 after inhalation of the provoking agent, indicating the presence of airway hyperresponsiveness. Bronchial provocation test can be performed when FEV1 is ≥70% of predicted value (excluding respiratory infections within 4 weeks). If FEV1 is <70% of predicted value, a bronchodilator test is prioritized.
3. Average daily diurnal variation in Peak Expiratory Flow (PEF) >10% (calculated as the sum of daily PEF diurnal variation for at least 7 consecutive days divided by the total number of days), excluding respiratory infections.

Cough severity score (CET) > 5 points. Patients previously diagnosed with CVA who discontinued inhaled medications for more than 3 months for any reason and now meet the above criteria.

Exclusion Criteria:

- Inability to cooperate with the diagnostic tests for asthma or uncooperative for other reasons.

Pregnancy. Comorbid severe diseases of other systems (e.g., cardiovascular, metabolic, immune, nervous, urinary, hematological) that may interfere with the normal conduct of this study.

A clear history of upper respiratory tract infection within the 4 weeks prior to enrollment.

History of alcohol abuse or substance abuse, or history of psychiatric illness, antagonistic personality, ulterior motives, paranoia, or other emotional or intellectual problems that may compromise the validity of informed consent or participation in the study.

Chest imaging indicates clinically significant abnormalities related to the symptoms.

Smoking: Defined as having smoked more than 100 cigarettes in one's lifetime and having smoked within the past 5 years. Otherwise, considered a non-smoker.

Current use of ACEI (Angiotensin-Converting Enzyme Inhibitor) medications. Concurrent participation in another drug clinical trial, or deemed unsuitable for inclusion in this study by the investigator for other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
symptom recurrence rate | 12 month follow up
  symptom recurrence rate in patients with cough variant asthma

IPD SHARING:
Plan to Share IPD: Yes